CLINICAL TRIAL: NCT00574249
Title: A Multi-center, Randomized, Vehicle-Controlled Study to Assess the Efficacy and Safety of Adalimumab in Combination With Topical Treatment (Calcipotriol/Betamethasone) in Subjects With Moderate to Severe Psoriasis and Insufficient Response to Classic Systemic Treatment (BELIEVE)
Brief Title: Adalimumab in Combination With Topical Treatment (Calcipotriol/Betamethasone) in Subjects With Moderate to Severe Psoriasis and Insufficient Response to Classic Systemic Treatment
Acronym: BELIEVE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Abbott (Industry)
Responsible Party: Marie Rosenfeld, Senior CRM, Abbott
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: M10-060
Record Dates: First submitted 2007-12-12; First posted 2007-12-17 (Estimated); Results first posted 2010-01-18 (Estimated); Last update posted 2011-04-13 (Estimated); Status verified 2011-04

CONDITIONS: Chronic Plaque Psoriasis
Keywords: Psoriasis; Moderate Psoriasis; Severe Psoriasis; Chronic Plaque Psoriasis; Severe Chronic Plaque Psoriasis
MeSH Terms: conditions — Psoriasis | interventions — Adalimumab; calcipotriene; betamethasone dipropionate, calcipotriol drug combination

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- adalimumab + placebo (Active Comparator): adalimumab + placebo (vehicle ointment)
  Interventions: Biological: adalimumab; Drug: placebo (vehicle ointment)
- adalimumab + calcipotriol/betamethasone (Active Comparator): adalimumab + calcipotriol/betamethasone ointment
  Interventions: Biological: adalimumab; Drug: Calcipotriol/Betamethasone Ointment

INTERVENTIONS:
Biological: adalimumab — subcutaneous injection using prefilled pen/syringe, solution containing 40 mg in 0.8 milliliters; 2 injections given at Baseline (Day 1) then once every other week from Weeks 1 though 15
  Other Names: ABT-D2E7; Humira
Drug: Calcipotriol/Betamethasone Ointment — Topical ointment (calcipotriol 50 mcg/g and betamethasone 500 mcg/g) to be applied once daily to affected psoriasis skin on trunk and extremities for first 4 weeks and as needed from Week 5 through Week 16
  Other Names: Daivobet
  Arms: adalimumab + calcipotriol/betamethasone
Drug: placebo (vehicle ointment) — Topical vehicle ointment (matching active calcipotriol/betamethasone ointment) to be applied once daily to affected psoriasis skin on trunk and extremities for first 4 weeks and as needed from Week 5 through Week 16
  Arms: adalimumab + placebo

SUMMARY:
The objective of this study is to assess the efficacy and safety of adalimumab in combination with topical psoriasis treatment, calcipotriol/betamethasone, vs. adalimumab in combination with matching vehicle in subjects with moderate to severe chronic plaque psoriasis.

DETAILED DESCRIPTION:
Additional information regarding sponsors: Abbott GmbH & Co. KG is sponsor for EU member states. Abbott US is sponsor for non-EU member states.

ELIGIBILITY:
Inclusion Criteria:

* Subject is >= 18 years of age
* Subject had a clinical diagnosis of chronic plaque psoriasis for at least 6 months, and has moderate to severe plaque psoriasis
* Subject must have been treated and failed to respond to, or has a contraindication to, or is intolerant to at least two different systemic therapies, one of which must be cyclosporine, or methotrexate or oral PUVA
* Subject is judged to be in generally good health as determined by the principal investigator

Exclusion Criteria:

* Subject has previous exposure to adalimumab
* Subject cannot discontinue systemic therapies and/or topical therapies for the treatment of psoriasis and cannot avoid UVB or PUVA phototherapy
* Subject is taking or requires oral or injectible corticosteroids
* Subject diagnosed with erythrodermic psoriasis, pustular psoriasis, medication-induced or medication-exacerbated psoriasis or new onset guttate psoriasis
* Subject considered by the investigator, for any reason, to be an unsuitable candidate
* Female subject who is pregnant or breast-feeding or considering becoming pregnant
* Subject has a calcium metabolism disorder

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 730 (Actual)
Dates: Start 2007-11; Primary Completion 2008-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (116):
- Austria (5):
  - Graz
  - Innsbruck
  - Salzburg
  - Vienna
  - Wein
- Belgium (10):
  - Aalst
  - Bruges
  - Brussels
  - Edegem
  - Geel
  - Ghent
  - Kortrijk
  - Leuven
  - Liège
  - Mons
- Czechia (3):
  - Brno
  - Hradec Králové
  - Prague
- Denmark (4):
  - Arhus C
  - Copenhagen
  - Hellerup
  - Herning
- Finland (3):
  - Helsinki HUS
  - Jyväskylä
  - Lahti
- France (13):
  - Brest
  - Créteil
  - Lille
  - Limoges
  - Montpellier
  - Nancy
  - Nice
  - Paris
  - Pessac
  - Pierre-Bénite
  - Rouen
  - Saint-Etienne
  - Toulouse
- Germany (26):
  - Berlin
  - Buchholz Nordheide
  - Cologne
  - Dresden
  - Düsseldorf
  - Erlangen
  - Frankfurt
  - Freiburg im Breisgau
  - Göttingen
  - Halle
  - Hamburg
  - Hanover
  - Heidelberg
  - Jena
  - Kiel
  - Leipzig
  - Magdeburg
  - Mainz
  - München
  - Münster
  - Oldenburg
  - Osnabrück
  - Potsdam
  - Regensburg
  - Rostock
  - Tübingen
- Greece (2):
  - Athens
  - Crete
- Italy (11):
  - Benevento
  - Catania
  - Catanzaro
  - Coppitto-L'Aquila
  - Florence
  - Messina
  - Milan
  - Modena
  - Padua
  - Palermo
  - Roma
- Netherlands (5):
  - Amsterdam
  - Breda
  - Maastricht
  - Nijmegen
  - Rotterdam
- Spain (14):
  - Alicante
  - Barcelona
  - Bilbao
  - Galdacano Vizcaya
  - Granada
  - Las Palmas de Gran Canarias
  - Madrid
  - Málaga
  - Santander
  - Santiago
  - Santiago de Compostela
  - Seville
  - Valencia
  - Vigo
- Sweden (4):
  - Falun
  - Gothenburg
  - Malmo
  - Stockholm
- Switzerland (4):
  - Basel
  - Bern
  - Geneva
  - Zurich
- Turkey (Türkiye) (4):
  - Ankara
  - Bursa
  - Çapa
  - Istanbul
- United Kingdom (8):
  - Aberdeen
  - Cardiff
  - Glasgow
  - Leeds
  - London
  - Manchester
  - Newport Gwent
  - Nuneaton

REFERENCES:
- [Derived] Paul C, van de Kerkhof P, Puig L, Unnebrink K, Goldblum O, Thaci D. Influence of psoriatic arthritis on the efficacy of adalimumab and on the treatment response of other markers of psoriasis burden: subanalysis of the BELIEVE study. Eur J Dermatol. 2012 Nov-Dec;22(6):762-9. doi: 10.1684/ejd.2012.1863. PMID 23178916

RESULTS

PARTICIPANT FLOW:
Groups:
- Adalimumab + Placebo: adalimumab + placebo (vehicle ointment): subcutaneous injection using prefilled pen/syringe, solution containing 40 mg adalimumab in 0.8 milliliters; 2 injections given at Baseline (Day 1) then one injection every other week from Week 1 through Week 15 - placebo vehicle ointment to be applied once daily to affected psoriasis skin on trunk and extremities for first 4 weeks and as needed from Week 5 though Week 16 (maximum dose of 100 g per week)
- Adalimumab + Calcipotriol/Betamethasone: adalimumab + calcipotriol/betamethasone ointment: subcutaneous injection using prefilled pen/syringe, solution containing 40 mg adalimumab in 0.8 milliliters; 2 injections given at Baseline (Day 1) then one injection every other week from Week 1 though Week 15 - topical ointment (calcipotriol 50 mcg/g and betamethasone 500 mg/g) to be applied once daily to affected psoriasis skin on trunk and extremities for first 4 weeks and as needed from Week 5 through Week 16 (maximum 100 g per week)
Period: Overall Study
Arm/Group | Adalimumab + Placebo | Adalimumab + Calcipotriol/Betamethasone
Started | 364 | 366
Completed | 338 | 338
Not Completed | 26 | 28
Not completed — Adverse Event | 6 | 18
Not completed — Lack of Efficacy | 5 | 3
Not completed — Lost to Follow-up | 4 | 3
Not completed — Protocol Violation | 5 | 2
Not completed — History of carcinoma | 1 | 0
Not completed — Withdrawal by Subject | 3 | 0
Not completed — Physician Decision | 1 | 0
Not completed — Pregnancy | 1 | 0
Not completed — Excluded by company | 0 | 1
Not completed — PPD test taken twice | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Adalimumab + Placebo: adalimumab + placebo (vehicle ointment): subcutaneous injection using prefilled pen/syringe, solution containing 40 mg adalimumab in 0.8 milliliters; 2 injections given at Baseline (Day 1) then one injection every other week from Week 1 through Week 15
- Total: Total of all reporting groups
Arm/Group | Adalimumab + Placebo | Adalimumab + Calcipotriol/Betamethasone | Total
Number analyzed (Participants) | 364 | 366 | 730
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 1 | 1
  Between 18 and 65 years | 343 | 350 | 693
  >=65 years | 21 | 15 | 36
Age Continuous [Mean (Standard Deviation); unit: years] | 44.8 (12.61) | 45.3 (11.95) | 45.1 (12.28)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 113 | 116 | 229
  Male | 251 | 250 | 501
Region of Enrollment [Number; unit: participants]
  Austria | 12 | 12 | 24
  Belgium | 40 | 36 | 76
  Czech Republic | 8 | 10 | 18
  Denmark | 15 | 15 | 30
  Finland | 5 | 6 | 11
  France | 58 | 61 | 119
  Germany | 79 | 83 | 162
  Greece | 12 | 12 | 24
  Italy | 32 | 34 | 66
  Netherlands | 17 | 18 | 35
  Spain | 33 | 26 | 59
  Sweden | 9 | 8 | 17
  Switzerland | 12 | 10 | 22
  Turkey | 14 | 14 | 28
  United Kingdom | 18 | 21 | 39

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Achieve a PASI75 Response at Week 16 Compared With Baseline (Week 0)
Description: PASI75 is defined as at least a 75% reduction in PASI (Psoriasis Area and Severity Index) score compared with the Baseline PASI score. PASI scores range from 0.0 (best) to 72.0 (worst), with the highest score representing complete erythroderma of the severest degree. The percent decrease in score is calculated as (Week 0 PASI score minus Week 16 PASI score) divided by Week 0 PASI score. Positive percent decreases indicate improvement, with best improvement being 100%. The outcome measure is the percentage of participants who had at least a 75% PASI score decrease.
Time Frame: Week 0 and Week 16
Population: ITT analysis; participants with a missing PASI assessment at Week 16 were imputed as nonresponders.
Measure: Number; unit: percentage of participants
Arm/Group | Adalimumab + Placebo | Adalimumab + Calcipotriol/Betamethasone
Number analyzed (Participants) | 364 | 366
percentage of participants | 70.9 | 64.8
Statistical Analysis 1: Comparison: Adalimumab + Placebo vs Adalimumab + Calcipotriol/Betamethasone; Comparison of the proportion of participants in the adalimumab + calcipotriol/betamethasone group vs. the adalimumab + placebo group; Test type: Superiority or Other; p = 0.086, Cochran-Mantel-Haenszel — Level of significance 5%; no adjustment for multiple comparisons necessary; Two-sided CMH test stratified by country at the alpha level 0.05. Centers were pooled by country (Sweden and Finland pooled due to few participants)

2. Secondary Outcome: Percentage of Participants With a PASI50 Response at Week 16 Compared With Baseline (Week 0)
Description: PASI50 is defined as at least a 50% reduction in PASI (Psoriasis Area and Severity Index) score compared with the Baseline PASI score. PASI scores range from 0.0 (best) to 72.0 (worst), with the highest score representing complete erythroderma of the severest degree. The percent decrease in score is calculated as (Week 0 PASI score minus Week 16 PASI score) divided by Week 0 PASI score. Positive percent decreases indicate improvement, with best improvement 100%. The outcome measure is the percentage of participants who had at least a 50% PASI score decrease.
Time Frame: Week 0 and Week 16
Population: ITT analysis; participants with a missing PASI assessment at Week 16 were imputed as nonresponders.
Measure: Number; unit: percentage of participants
Arm/Group | Adalimumab + Placebo | Adalimumab + Calcipotriol/Betamethasone
Number analyzed (Participants) | 364 | 366
percentage of participants | 82.7 | 80.9
Statistical Analysis 1: Comparison: Adalimumab + Placebo vs Adalimumab + Calcipotriol/Betamethasone; Test type: Superiority or Other; p = 0.565, Fisher Exact

3. Secondary Outcome: Percentage of Participants With a PASI90 Response at Week 16 Compared With Baseline (Week 0)
Description: PASI90 is defined as at least a 90% reduction in PASI (Psoriasis Area and Severity Index) score compared with the Baseline PASI score. PASI scores range from 0.0 (best) to 72.0 (worst), with the highest score representing complete erythroderma of the severest degree. The percent decrease in score is calculated as (Week 0 PASI score minus Week 16 PASI score) divided by Week 0 PASI score. Positive percent decreases indicate improvement, with best improvement 100%. The outcome measure is the percentage of participants who had at least a 90% PASI score decrease.
Time Frame: Week 0 and Week 16
Population: ITT analysis; participants with a missing PASI assessment at Week 16 were imputed as nonresponders.
Measure: Number; unit: percentage of participants
Arm/Group | Adalimumab + Placebo | Adalimumab + Calcipotriol/Betamethasone
Number analyzed (Participants) | 364 | 366
percentage of participants | 50.3 | 38.8
Statistical Analysis 1: Comparison: Adalimumab + Placebo vs Adalimumab + Calcipotriol/Betamethasone; Test type: Superiority or Other; p = 0.002, Fisher Exact

4. Secondary Outcome: Percentage of Participants With a PASI100 Response at Week 16 Compared With Baseline (Week 0)
Description: PASI100 is defined as at least a 100% reduction in PASI (Psoriasis Area and Severity Index) score compared with the Baseline PASI score. PASI scores range from 0.0 (best) to 72.0 (worst) with the highest score representing complete erythroderma of the severest degree. The percent decrease in score is calculated as (Week 0 PASI score minus Week 16 PASI score) divided by Week 0 PASI score. Positive percent decreases indicate improvement, with best improvement 100%. The outcome measure is the percentage of participants who had at least a 100% PASI score decrease.
Time Frame: Week 0 and Week 16
Population: ITT analysis; participants with a missing PASI assessment at Week 16 were imputed as nonresponders.
Measure: Number; unit: percentage of participants
Arm/Group | Adalimumab + Placebo | Adalimumab + Calcipotriol/Betamethasone
Number analyzed (Participants) | 364 | 366
percentage of participants | 24.2 | 15.3
Statistical Analysis 1: Comparison: Adalimumab + Placebo vs Adalimumab + Calcipotriol/Betamethasone; Test type: Superiority or Other; p = 0.003, Fisher Exact

5. Secondary Outcome: Percentage of Participants Achieving a Physician's Global Assessment (PGA) of Clear or Minimal at Week 2
Description: PGA is a physician's assessment of severity of disease (grading lesion severity). PGA scores range from 0 (best) to 6 (worst): on the 6-point scale, a score of 0 = Clear and a score of 6 = Very Severe for the lesion severity. PGA Clear (0) is no plaque elevation over normal skin and no scale with or without erythema. Minimal (1) is possible plaque elevation but difficult to ascertain a slight elevation above normal skin. Percentage of participants: 0% to 100% (best).
Time Frame: Week 2
Population: ITT analysis. Imputation of missing values at Week 2 as not achieving PGA of Clear or Minimal.
Measure: Number; unit: percentage of participants
Arm/Group | Adalimumab + Placebo | Adalimumab + Calcipotriol/Betamethasone
Number analyzed (Participants) | 364 | 366
percentage of participants | 7.1 | 13.9
Statistical Analysis 1: Comparison: Adalimumab + Placebo vs Adalimumab + Calcipotriol/Betamethasone; Test type: Superiority or Other; p = 0.004, Fisher Exact

6. Secondary Outcome: Percentage of Participants Achieving a Physician's Global Assessment (PGA) of Clear or Minimal at Week 4
Description: as for outcome 5
Time Frame: Week 4
Population: ITT analysis. Imputation of missing values at Week 4 as not achieving PGA of Clear or Minimal.
Measure: Number; unit: percentage of participants
Arm/Group | Adalimumab + Placebo | Adalimumab + Calcipotriol/Betamethasone
Number analyzed (Participants) | 364 | 366
percentage of participants | 24.5 | 33.1
Statistical Analysis 1: Comparison: Adalimumab + Placebo vs Adalimumab + Calcipotriol/Betamethasone; Test type: Superiority or Other; p = 0.011, Fisher Exact

7. Other Pre Specified Outcome: Percent Change in Psoriasis Scalp Severity Index (PSSI) From Baseline to Week 16.
Description: PSSI is a physician assessment of clinical symptoms of scalp psoriasis. Computed as the sum of scores for erythema, induration, and desquamation (1 = absent; 4 = severest possible) multiplied by involved area (0 = 0%; 6 = 90-100%). Total score range: 0 (best) to 72 (worst). Negative change and percent change from Baseline indicate improvement.
Time Frame: Week 0 and Week 16
Population: Of the ITT analysis set, participants with a PSSI score at both Baseline and Week 16. Imputation of missing values using LOCF. Subjects with a zero score at Baseline were not included in analysis of percent change.
Measure: Median (Inter-Quartile Range); unit: percent change in score
Arm/Group | Adalimumab + Placebo | Adalimumab + Calcipotriol/Betamethasone
Number analyzed (Participants) | 321 | 319
percent change in score | -100.00 [-100.0 to -87.5] | -100.00 [-100.0 to -80.0]
Statistical Analysis 1: Comparison: Adalimumab + Placebo vs Adalimumab + Calcipotriol/Betamethasone; Test type: Superiority or Other; p = 0.204, ANOVA; One-way ANOVA. For confidence interval and difference estimate, adalimumab + calcipotriol/betamethasone minus adalimumab + placebo was used; Mean Difference (Net) = 9.74, 95% CI [-5.30 to 24.78]

8. Other Pre Specified Outcome: Percent Change in Nail Psoriasis Severity Index (NAPSI) at Week 16.
Description: NAPSI is a sum of 2 scores that grade nail matrix psoriasis (based on presence/absence of pitting, leukonychia, red spots in the lunula, and nail plate crumbling) and nail bed psoriasis (based on presence/absence of onycholysis splinter hemorrhages, oil drop [salmon patch] discoloration, and nail bed hyperkeratosis). Each fingernail is given a single score based on presence of psoriasis in quadrant of nail: 0 (none) to 4 (present in 4/4 nail quadrants). Score range: 0 (best) to 80 (worst). Negative change and percent change from Baseline indicate improvement.
Time Frame: Week 0 and Week 16
Population: Of the ITT analysis set, participants with a NAPSI score at both Baseline and Week 16. Imputation of missing values using LOCF. Subjects with a zero score at Baseline were not included in analysis of percent change.
Measure: Median (Inter-Quartile Range); unit: percent change in score
Arm/Group | Adalimumab + Placebo | Adalimumab + Calcipotriol/Betamethasone
Number analyzed (Participants) | 213 | 212
percent change in score | -40.00 [-66.7 to 0.0] | -37.50 [-68.4 to 0.0]
Statistical Analysis 1: Comparison: Adalimumab + Placebo vs Adalimumab + Calcipotriol/Betamethasone; Test type: Superiority or Other; p = 0.272, ANOVA; One-way ANOVA. Confidence interval and difference estimated from adalimumab + calcipotriol/betamethasone minus adalimumab + placebo; Mean Difference (Net) = -17.55, 95% CI [-48.92 to 13.82]

9. Secondary Outcome: Percentage of Participants Achieving a Physician's Global Assessment (PGA) of Clear or Minimal at Week 8
Description: as for outcome 5
Time Frame: Week 8
Population: ITT analysis. Imputation of missing values at Week 8 as not achieving PGA of Clear or Minimal.
Measure: Number; unit: percentage of participants
Arm/Group | Adalimumab + Placebo | Adalimumab + Calcipotriol/Betamethasone
Number analyzed (Participants) | 364 | 366
percentage of participants | 46.2 | 42.9
Statistical Analysis 1: Comparison: Adalimumab + Placebo vs Adalimumab + Calcipotriol/Betamethasone; Test type: Superiority or Other; p = 0.413, Fisher Exact

10. Secondary Outcome: Percentage of Participants Achieving a Physician's Global Assessment (PGA) of Clear or Minimal at Week 12
Description: as for outcome 5
Time Frame: Week 12
Population: ITT analysis. Imputation of missing values at Week 12 as not achieving PGA of Clear or Minimal.
Measure: Number; unit: percentage of participants
Arm/Group | Adalimumab + Placebo | Adalimumab + Calcipotriol/Betamethasone
Number analyzed (Participants) | 364 | 366
percentage of participants | 64.8 | 50.0
Statistical Analysis 1: Comparison: Adalimumab + Placebo vs Adalimumab + Calcipotriol/Betamethasone; Test type: Superiority or Other; p < 0.001, Fisher Exact

11. Secondary Outcome: Percentage of Participants Achieving a Physicians Global Assessment (PGA) Response of Clear or Minimal at Week 16
Description: as for outcome 5
Time Frame: Week 16
Population: ITT analysis. Imputation of missing values at Week 16 as not achieving PGA of Clear or Minimal.
Measure: Number; unit: percentage of participants
Arm/Group | Adalimumab + Placebo | Adalimumab + Calcipotriol/Betamethasone
Number analyzed (Participants) | 364 | 366
percentage of participants | 64.6 | 56.6
Statistical Analysis 1: Comparison: Adalimumab + Placebo vs Adalimumab + Calcipotriol/Betamethasone; Test type: Superiority or Other; p = 0.028, Fisher Exact

12. Secondary Outcome: Percent Change From Baseline in the Dermatology Life Quality Index (DLQI) Total Score at Week 16 Compared With Baseline (Week 0)
Description: DLQI is a participant-reported outcome consisting of a set of 10 questions regarding the degree to which (i.e., how much) the subject's skin has affected certain behaviors and quality of life over the last week. Responses to each are: very much, a lot, a little, or not at all. Total score range: 0 (best) to 30 (worst). Negative change and percent change from Baseline indicate improvement, with best improvement -100%.
Time Frame: Week 0 and Week 16
Population: Of the ITT analysis set, participants with DLQI scores both at Baseline and Week 16. Imputation of missing values using last observation carried forward (LOCF). Participants with a zero score at Baseline were not included in analysis of percent change.
Measure: Mean (Standard Deviation); unit: percent change in score
Arm/Group | Adalimumab + Placebo | Adalimumab + Calcipotriol/Betamethasone
Number analyzed (Participants) | 354 | 363
percent change in score | -71.46 (49.171) | -67.20 (45.463)
Statistical Analysis 1: Comparison: Adalimumab + Placebo vs Adalimumab + Calcipotriol/Betamethasone; Test type: Superiority or Other; p = 0.228, ANOVA; One-way ANOVA

13. Secondary Outcome: Percent Change in the Dermatology Life Quality Index (DLQI) Total Score at Week 2 Compared With Baseline (Week 0)
Description: as for outcome 12
Time Frame: Week 0 and Week 2
Population: Of the ITT analysis set, participants with DLQI scores at both Baseline and Week 2. Imputation of missing values using LOCF. Participants with a zero score at Baseline were not included in analysis of percent change.
Measure: Mean (Standard Deviation); unit: percent change in score
Arm/Group | Adalimumab + Placebo | Adalimumab + Calcipotriol/Betamethasone
Number analyzed (Participants) | 346 | 361
percent change in score | -32.14 (44.118) | -47.49 (41.093)
Statistical Analysis 1: Comparison: Adalimumab + Placebo vs Adalimumab + Calcipotriol/Betamethasone; Test type: Superiority or Other; p < 0.001, ANOVA; One-way ANOVA

14. Secondary Outcome: Percent Change From Baseline in the Dermatology Life Quality Index (DLQI) Total Score at Week 4 Compared With Baseline (Week 0)
Description: as for outcome 12
Time Frame: Week 0 and Week 4
Population: Of the ITT analysis set, participants with DLQI scores at both Baseline and Week 4. Imputation of missing values using LOCF. Participants with a zero score at Baseline were not included in the analysis of percent change.
Measure: Mean (Standard Deviation); unit: percent change in score
Arm/Group | Adalimumab + Placebo | Adalimumab + Calcipotriol/Betamethasone
Number analyzed (Participants) | 354 | 362
percent change in score | -46.64 (68.139) | -60.93 (38.122)
Statistical Analysis 1: Comparison: Adalimumab + Placebo vs Adalimumab + Calcipotriol/Betamethasone; Test type: Superiority or Other; p = 0.001, ANOVA; One-way ANOVA

15. Secondary Outcome: Percent Change From Baseline in the Dermatology Life Quality Index (DLQI) Total Score at Week 8 Compared With Baseline (Week 0)
Description: as for outcome 12
Time Frame: Week 0 and Week 8
Population: Of the ITT analysis set, participants with DLQI scores at both Baseline and Week 8. Imputation of missing values using LOCF. Participants with a zero score at Baseline were not included in analysis of percent change.
Measure: Mean (Standard Deviation); unit: percent change in score
Arm/Group | Adalimumab + Placebo | Adalimumab + Calcipotriol/Betamethasone
Number analyzed (Participants) | 354 | 363
percent change in score | -63.30 (45.404) | -62.30 (43.087)
Statistical Analysis 1: Comparison: Adalimumab + Placebo vs Adalimumab + Calcipotriol/Betamethasone; Test type: Superiority or Other; p = 0.764, ANOVA; One-way ANOVA

16. Secondary Outcome: Percent Change From Baseline in the Dermatology Life Quality Index (DLQI) Total Score at Week 12 Compared With Baseline (Week 0)
Description: as for outcome 12
Time Frame: Week 0 and Week 12
Population: Of the ITT analysis set, participants with DLQI scores at both Baseline and Week 12. Imputation of missing values using LOCF. Participants with a zero score at Baseline were not included in analysis of percent change.
Measure: Mean (Standard Deviation); unit: percent change in score
Arm/Group | Adalimumab + Placebo | Adalimumab + Calcipotriol/Betamethasone
Number analyzed (Participants) | 354 | 363
percent change in score | -69.49 (45.030) | -66.75 (49.195)
Statistical Analysis 1: Comparison: Adalimumab + Placebo vs Adalimumab + Calcipotriol/Betamethasone; Test type: Superiority or Other; p = 0.437, ANOVA; One-way ANOVA

17. Secondary Outcome: Percent Change in Short Form 36 Health Survey (SF-36) Physical Component Score (PCS) at Week 16 Compared With Baseline (Week 0)
Description: Short Form 36 Health Survey (SF-36) Physical Component Score (PCS) is a participant-reported outcome that employs a questionnaire that asks for the participant's views about their health. Percent change at Week 16 is calculated as (Week 16 SF-36 PCS minus Week 0 SF-36 PCS) divided by Week 0 SF-36 PCS. Positive percent change in score indicates improvement, with best improvement 100%.
Time Frame: Week 0 and Week 16
Population: Of the ITT analysis set, participants with an SF-36 score at both Baseline and Week 16. Imputation of missing values using LOCF. Participants with a zero score at Baseline were not included in the analysis of percent change.
Measure: Mean (Standard Deviation); unit: percent change in score
Arm/Group | Adalimumab + Placebo | Adalimumab + Calcipotriol/Betamethasone
Number analyzed (Participants) | 333 | 333
percent change in score | 20.53 (31.603) | 19.71 (32.136)
Statistical Analysis 1: Comparison: Adalimumab + Placebo vs Adalimumab + Calcipotriol/Betamethasone; Test type: Superiority or Other; p = 0.740, ANOVA; One-way ANOVA

18. Secondary Outcome: Percent Change in Short Form 36 Health Survey (SF-36) Physical Component Score (PCS) at Week 8 Compared With Baseline (Week 0)
Description: Short Form 36 Health Survey (SF-36) Physical Component Score (PCS) is a participant-reported outcome that employs a questionnaire that asks for the participant's views about their health. Percent change at Week 8 is calculated as (Week 8 SF-36 PCS minus Week 0 SF-36 PCS) divided by Week 0 SF-36 PCS. Positive percent change in score indicates improvement, with best improvement 100%.
Time Frame: Week 0 and Week 8
Population: Of the ITT analysis set, participants with an SF-36 score both at Baseline and Week 8. Imputation of missing values using LOCF. Participants with a zero score at Baseline were not included in the analysis of percent change.
Measure: Mean (Standard Deviation); unit: percent change in score
Arm/Group | Adalimumab + Placebo | Adalimumab + Calcipotriol/Betamethasone
Number analyzed (Participants) | 327 | 321
percent change in score | 19.35 (30.264) | 18.22 (29.967)
Statistical Analysis 1: Comparison: Adalimumab + Placebo vs Adalimumab + Calcipotriol/Betamethasone; Test type: Superiority or Other; p = 0.634, ANOVA; One-way ANOVA

ADVERSE EVENTS:
Time Frame: Overall study
Arm/Group | Adalimumab + Placebo | Adalimumab + Calcipotriol/Betamethasone
Serious Adverse Events (participants affected / at risk) | 15/364 | 16/366
Other Adverse Events (participants affected / at risk) | 124/364 | 136/366
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Adalimumab + Placebo (N=364) | Adalimumab + Calcipotriol/Betamethasone (N=366)
angina pectoris (Cardiac disorders) | 1 | 0
retinal vein thrombosis (Eye disorders) | 0 | 1
vitreous haemorrhage (Eye disorders) | 0 | 1
oedema peripheral (General disorders) | 0 | 1
hepatitis (Hepatobiliary disorders) | 0 | 1
anaphylatic shock (Immune system disorders) | 1 | 0
abortion infected (Infections and infestations) | 1/113 | 0/116
bronchopneumonia (Infections and infestations) | 1 | 0
erysipelas (Infections and infestations) | 1 | 1
herpes zoster (Infections and infestations) | 0 | 1
localised infection (Infections and infestations) | 0 | 1
osteomyelitis (Infections and infestations) | 0 | 1
pneumonia (Infections and infestations) | 0 | 2
staphylococcal infection (Infections and infestations) | 1 | 0
arteriogram coronary (Investigations) | 0 | 1
joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 1
musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0
pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1
lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
rectal adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
convulsion (Nervous system disorders) | 1 | 0
acute generalised exanthematous pustulosis (Skin and subcutaneous tissue disorders) | 1 | 0
dermatitis exfoliative (Skin and subcutaneous tissue disorders) | 2 | 0
dry skin (Skin and subcutaneous tissue disorders) | 1 | 0
onycholysis (Skin and subcutaneous tissue disorders) | 0 | 1
psoriasis (Skin and subcutaneous tissue disorders) | 1 | 1
skin inflammation (Skin and subcutaneous tissue disorders) | 1 | 0
peripheral vascular disorder (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Adalimumab + Placebo (N=364) | Adalimumab + Calcipotriol/Betamethasone (N=366)
Diarrhoea (Gastrointestinal disorders) | 7 | 11
Nausea (Gastrointestinal disorders) | 5 | 12
Asthenia (General disorders) | 2 | 8
Fatigue (General disorders) | 9 | 8
Injection site pain (General disorders) | 8 | 3
Influenza (Infections and infestations) | 8 | 6
Nasopharyngitis (Infections and infestations) | 23 | 32
Oral herpes (Infections and infestations) | 6 | 9
Rhinitis (Infections and infestations) | 10 | 4
Arthralgia (Musculoskeletal and connective tissue disorders) | 7 | 11
Headache (Nervous system disorders) | 22 | 19
Cough (Respiratory, thoracic and mediastinal disorders) | 12 | 11
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 8 | 9
Pruritus (Skin and subcutaneous tissue disorders) | 21 | 13
Psoriasis (Skin and subcutaneous tissue disorders) | 17 | 19
Hypertension (Vascular disorders) | 4 | 10
Pharyngitis (Infections and infestations) | 12 | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Investigator shall provide Abbott at least (60) days prior to publication or presentation, for Abbott's review and comment, to ascertain whether any patent subject matter or Abbott confidential information are disclosed. During the review, Abbott may request a delay for up to six (6) months from the date of first submission to Abbott in order to protect proprietary information.